CLINICAL TRIAL: NCT01565668
Title: A Phase 2, Randomized, Open-Label Study of the Safety and Efficacy of Two Doses of Quizartinib (AC220; ASP2689) in Subjects With FLT3-ITD Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Open Label Study to Evaluate Safety and Efficacy of 2 Doses of Quizartinib in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Ambit Biosciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2689-CL-2004; 2011-005408-13 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: FLT3-ITD positive Acute Myeloid Leukemia (AML); AC220; Relapse; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC220 Dose Level 1 (Experimental)
  Interventions: Drug: AC220
- AC220 Dose Level 2 (Experimental)
  Interventions: Drug: AC220

INTERVENTIONS:
Drug: AC220 — oral
  Other Names: Quizartinib; ASP2689

SUMMARY:
This study will evaluate two doses of Quizartinib in patients with relapsed or refractory acute myeloid leukemia who are also FMS-like tyrosine kinase - internal tandem duplication ( FLT3-ITD) positive. Patient will be randomly assigned in a 1:1 ratio to one of two treatment arms. Both treatment arms will receive Quizartinib but at different doses. The study treatment is taken orally in 28 day cycles until either disease progression occurs or an unacceptable toxicity occurs. In addition to the study assessments to evaluate the disease, blood will be drawn to measure drug levels and biomarkers. Patients will be followed for survival at three month intervals after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has morphologically documented primary acute myeloid leukemia (AML) or AML secondary to myelodysplastic syndrome (MDS) as defined by the World Health Organization (WHO) criteria, as determined by pathology review at the treating institution and has relapsed or is refractory after 1 second line (salvage) regimen or after hematopoietic stem cell transplantation (HSCT)
* Subject is positive for FLT3-ITD activating mutation in bone marrow or peripheral blood (>10% allelic ratio)
* Eastern Cooperative Oncology Group performance status of 0 to 2
* In the absence of rapidly progressing disease clearly documented by the investigator, the interval from prior treatment to time of AC220 administration will be at least 2 weeks (14 days) for prior cytotoxic agents or at least 5 half-lives for prior noncytotoxic agents, including immunosuppressive therapy post HSCT
* Persistent chronic clinically significant nonhematological toxicities from prior treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation, HSCT, or surgery) must be Grade ≤ 1
* Patients - both males and females - with reproductive potential are eligible

Exclusion Criteria:

* Subject received previous treatment with AC220
* Subject has a diagnosis of acute promyelocytic leukemia
* Subject has a diagnosis of chronic myelogenous leukemia (CML) in blast crisis
* Subject has AML or antecedent MDS secondary to prior chemotherapy
* Subject has had HSCT and has either of the following:
* Donor lymphocyte infusion (DLI) is not permitted during the study or < 30 days prior to study entry
* Subject has clinically active central nervous system (CNS) leukemia. A subject is considered eligible if CNS leukemia is controlled and subject is receiving intrathecal (IT) therapy at study entry. Subjects should continue to receive IT therapy (or cranial radiation) as clinically indicated
* Subject has received concurrent chemotherapy, immunotherapy, or radiotherapy within 14 days prior to the first dose of AC220, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation) within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
* Subject requires treatment with concomitant drugs that prolong QT/QTc interval or with strong inhibitors or inducers of cytochrome P450- isozyme3A4 (CYP3A4) with the exception of antibiotics, antifungals, and antivirals that are used as standard of care post-transplant or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject
* Subject requires treatment with anticoagulant therapy
* Subject has a known positive test for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen
* Subject had major surgery within 4 weeks prior to first dose of AC220
* Subject has uncontrolled or significant cardiovascular disease, including
* Subject has a pre-existing disorder predisposing the subject to a serious or life-threatening infection (e.g. cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias not related to AML)
* Subject has an active uncontrolled acute or chronic systemic fungal, bacterial, viral, or other infection
* Subject has any of the following laboratory values:
* Subject is a female with a positive pregnancy test, pregnant, or breastfeeding
* Subject has any medical, psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (24):
- United States (18):
  - UCLA School of Medicine, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - John Hopkins University, Baltimore, Maryland
  - Tufts University School of Medicine-Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University, Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Simmons Cancer Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (4):
  - CHU d'Angers, Angers
  - CHU de Grenoble, Grenoble
  - Hôpital Saint Antoine, Paris
  - Hôpital Haut Lévêque, Pessac
- Universitaria Policlinico S. Orsola Malpighi, Institute of Hemtology "L. & A. Seragnoli", Bologna, Italy
- Nottingham University Hospitals, Nottingham, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 76 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study (intent-to-treat population). Participants were enrolled at 22 clinic sites in North America and Europe (14 sites in the United States, 6 in France, 1 in Italy, and 1 in the United Kingdom).
Pre-assignment Details: Participants were randomized (1:1) to receive 30 or 60 mg/day quizartinib. These doses were selected based on evidence of efficacy and safety observed in studies AC220-001 and AC220-002, and preclinical data.Two participants who were randomized to quizartinib (60 mg/day) did not receive study drug and are not included in the safety data.
Groups:
- Quizartinib 30 mg: Participants randomized to receive 30 mg quizartinib once daily.
- Quizartinib 60 mg: Participants randomized to receive 60 mg quizartinib once daily.
Period: Overall Study
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Started | 38 | 38
Completed Treatment Per Protocol | 0 | 0
Started 30-day Follow-up | 37 | 37
Completed 30-day Follow-up | 11 | 5
Started Long-term Follow-up | 36 | 33
Completed Long-term Follow-up | 0 | 0
Completed | 0 | 0
Not Completed | 38 | 38
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 4 | 2
Not completed — Participant went on Hospice Care | 1 | 0
Not completed — Adverse Event | 6 | 1
Not completed — Randomized, but never received drug | 0 | 2
Not completed — Progressive disease | 13 | 14
Not completed — Withdrawal by Subject | 1 | 3
Not completed — HSCT Transplant | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Quizartinib 60 mg: Participants were randomized to receive 60 mg quizartinib once daily.
- Total: Total of all reporting groups
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Median (Full Range); unit: years] | 56.5 [19 to 77] | 53.0 [20 to 74] | 54.5 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
  Italy | 0 | 3 | 3
  United Kingdom | 2 | 1 | 3
  France | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Composite Complete Response (CRc) (Intent-to-Treat Population)
Description: CRc is defined as Complete remission (CR) + Complete remission with incomplete platelet recovery (CRp) + Complete remission with incomplete hematological recovery (CRi).
  * Participants with CR must have normal hematopoietic cells and achieved a morphologic leukemia-free state (<5% bone marrow blasts in bone marrow, no blasts with Auer rods and no persistence of extramedullary disease) and must have had an absolute neutrophil count (ANC) ≥1 × 10^9/L and platelet count ≥100 × 10^9/L and were red blood cell (RBC) and platelet transfusion independent. Blasts in the peripheral blood was to be ≤1% (if blood sample was available).
  * Participants with CRp must have achieved CR except for incomplete platelet recovery (< 100 ×10^9/L).
  * Participants with CRi must have fulfilled all the criteria for CR except for incomplete hematological recovery with residual neutropenia <1 × 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence were not required.
Time Frame: At end of Cycle 2 (after two complete 28-day cycles post treatment)
Population: Composite complete remission was assessed in the intent-to-treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
Participants | 18 | 18

2. Secondary Outcome: Number of Participants Who Achieved Complete Remission (CR) (Intent-to-Treat Population)
Description: Participant must have bone marrow regenerating normal hematopoietic cells and achieve a morphologic leukemia-free state (< 5% bone marrow blasts in bone marrow, no blasts with Auer rods and no persistence of extramedullary disease) and must have an absolute neutrophil count (ANC) ≥ 1x10^9/L and platelet count ≥ 100 x 10^9/L and they will be red blood cell (RBC) and platelet transfusion independent (defined as 4 weeks without RBC transfusions and 1 week without platelet transfusion).
Time Frame: At end of treatment visit (approximately 3 years post treatment)
Population: Complete remission was assessed in the intent-to-treat (ITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
Participants | 2 | 1

3. Secondary Outcome: Overall Survival (OS) After Approximately 3 Years (Intent-to-Treat Population)
Description: OS was defined as the time from the date of randomization until the date of death from any cause.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: OS was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
weeks | 20.9 [17.7 to 25.3] | 27.3 [17.3 to 34.9]

4. Secondary Outcome: Event Free Survival (EFS) After Approximately 3 Years (Intent-to-Treat Population)
Description: EFS was defined as the time from the date of randomization until the date of documented relapse or death.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: EFS was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
weeks | 12.0 [8.3 to 16.1] | 13.7 [9.7 to 26.1]

5. Secondary Outcome: Leukemia Free Survival (LFS) After Approximately 3 Years (Intent-to-Treat Population)
Description: LFS was defined as the time from the date of first CRc until the date of documented relapse or death for participants who achieved CRc.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: LFS was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 18 | 18
weeks | 4.1 [2.1 to 9.7] | 9.1 [4.0 to 22.3]

6. Secondary Outcome: Duration of Remission After Approximately 3 Years (Intent-to-Treat Population)
Description: Duration of remission was defined as the time from first documented remission until documented relapse. CRc was defined as composite complete remission and CRi was defined as complete remission with incomplete hematological recovery.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: Duration of remission was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
weeks
  CRc: number analyzed (Participants) | 18 | 18
  CRc | 4.2 [2.1 to 9.7] | 9.1 [4.1 to 22.3]
  CRi: number analyzed (Participants) | 16 | 17
  CRi | 4.1 [2.1 to 9.7] | 20.0 [4.0 to 75.6]

7. Secondary Outcome: Time to Composite Complete Remission (CRc) in Participants Who Achieved CRc After Approximately 3 Years (Intent-to-Treat Population)
Description: Time to CRc was defined as the time from the date of randomization until the first disease assessment of CRc. Time to CRc was only evaluated in participants who achieved CRc.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: Time to CRc was assessed in the intent-to-treat (ITT) analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 18 | 18
weeks | 4.4 [4.1 to 7.7] | 4.6 [4.1 to 8.0]

8. Secondary Outcome: Percentage of Participants Undergoing Hematopoietic Stem Cell Transplantation (HSCT) After Approximately 3 Years (Intent-to-Treat Population)
Description: Transplantation rate was defined as the percentage of participants who underwent HSCT directly after treatment with quizartinib (no other intervening acute myeloid leukemia therapies other than conditioning regimens for the HSCT).
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: Transplantation rate was assessed in the intent-to-treat (ITT) analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 38
percentage of participants
  Yes | 31.6 | 42.1
  No | 68.4 | 55.3
  Unknown | 0 | 2.6

9. Secondary Outcome: Percentage of Participants With Grade 2 or Higher QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) Prolongation After Receiving Quizartinib (Safety Analysis Set)
Description: QT interval corrected for heart rate using Fridericia's formula (QTcF) grading was to be done according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and the definition of Grade 2 or higher prolongation is QTcF more than 480 msec.
Time Frame: Evaluated at end of study, up to 6 months (approximately 3 years post treatment)
Population: QTcF prolongation was assessed in the Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
Number analyzed (Participants) | 38 | 36
percentage of participants
  Max on study; <450 msec | 47.4 | 36.1
  Max on study; ≥450 msec and ≤480 msec | 42.1 | 47.2
  Max on study; >480 msec and ≤500 msec | 5.3 | 13.9
  Max on study; >500 msec | 5.3 | 2.8
  Max change from baseline; ≤30 msec | 47.4 | 38.9
  Max change from baseline; >30 msec and ≤60 msec | 47.4 | 41.7
  Max change from baseline; >60 msec | 5.3 | 19.4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first dose of treatment up to 30 days from the last dose of treatment in the safety analysis set. Two participants in the quizartinib 60 mg cohort did not receive the study drug and were not included in the safety analysis set.
Arm/Group | Quizartinib 30 mg | Quizartinib 60 mg
All-Cause Mortality (participants affected / at risk) | 9/38 | 13/36
Serious Adverse Events (participants affected / at risk) | 25/38 | 23/36
Other Adverse Events (participants affected / at risk) | 37/38 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 30 mg (N=38) | Quizartinib 60 mg (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 5
Multi-organ failure (General disorders) | 0 | 2
Pneumonia (Infections and infestations) | 3 | 6
Cellulitis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 2
Device-related infection (Infections and infestations) | 2 | 0
Periorbital cellulitis (Infections and infestations) | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Renal failure acute (Renal and urinary disorders) | 0 | 2
Urinary rentention (Renal and urinary disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Cecitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 1
Disease progression (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Bronchitis fungal (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Catheter-site infection (Infections and infestations) | 0 | 1
Clostridium difficile sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Klebsiella bacteremia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Medical observation (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Shock hemorrhagic (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quizartinib 30 mg (N=38) | Quizartinib 60 mg (N=36)
Anemia (Blood and lymphatic system disorders) | 18 | 9
Nausea (Gastrointestinal disorders) | 10 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 13
Pyrexia (General disorders) | 11 | 14
Vomiting (Gastrointestinal disorders) | 11 | 13
Diarrhea (Gastrointestinal disorders) | 10 | 13
Fatigue (General disorders) | 13 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Abdominal pain (Gastrointestinal disorders) | 6 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 7
Hypokalemia (Metabolism and nutrition disorders) | 9 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Oedema peripheral (General disorders) | 8 | 6
Headache (Nervous system disorders) | 4 | 9
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Mucosal inflammation (General disorders) | 6 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumonia (Infections and infestations) | 3 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hypotension (Vascular disorders) | 6 | 4
Tachycardia (Cardiac disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 6 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 4
Alanine aminotransferase increased (Investigations) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Chills (General disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Blood bilirubin increased (Investigations) | 3 | 4
Dizziness (Nervous system disorders) | 3 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 2 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Anxiety (Psychiatric disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 4
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Pain (General disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Asthenia (General disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Hemorrhoids (Gastrointestinal disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Non-cardiac chest pain (General disorders) | 0 | 5
Pericardial effusion (Cardiac disorders) | 3 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 2
Cellulitis (Infections and infestations) | 1 | 3
Clostridial infection (Infections and infestations) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oedema (General disorders) | 1 | 3
Paresthesia (Nervous system disorders) | 1 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 3
Platelet count decreased (Investigations) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Vision blurred (Eye disorders) | 3 | 1
Catheter site erythema (General disorders) | 1 | 2
Catheter site pain (General disorders) | 2 | 1
Chest discomfort (General disorders) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 1
Hematemesis (Gastrointestinal disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Herpes simplex (Infections and infestations) | 1 | 2
Melaena (Gastrointestinal disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 3
Rhinitis (Infections and infestations) | 1 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Septic shock (Infections and infestations) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 1
Tremor (Nervous system disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2
White blood cell count decreased (Investigations) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Ageusia (Nervous system disorders) | 0 | 2
Bacteremia (Infections and infestations) | 2 | 0
Blood alkaline phophatase increased (Investigations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Eructation (Gastrointestinal disorders) | 2 | 0
Escherichia sepsis (Infections and infestations) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Mouth hemorrhage (Gastrointestinal disorders) | 0 | 2
Multi-organ failure (General disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 2
Periorbital cellulitis (Infections and infestations) | 2 | 0
Pneumonia fungal (Infections and infestations) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary hesitation (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No